CLINICAL TRIAL: NCT01511731
Title: Open-label, Randomized, 2-way Crossover Study to Compare the Bioavailability of Reddy Cheminor and Merck &Co, Pepcid Famotidine Tablets 40 mg Under Fasting Conditions.
Brief Title: Bioavailability Study of Famotidine Tablets 40 mg Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 981325
Record Dates: First submitted 2012-01-12; First posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: Bioequivalence; famotidine; Crossover
MeSH Terms: interventions — Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Famotidine (Experimental): Famotidine tablets 40 mg of Dr. Reddy's
  Interventions: Drug: Famotidine
- Pepcid (Active Comparator): Pepcid 40 mg Tablets of Merck & Co.,
  Interventions: Drug: Pepcid

INTERVENTIONS:
Drug: Famotidine — Famotidine Tablets 40 mg
  Other Names: Reddy Cheminor
  Arms: Famotidine
Drug: Pepcid — 40mg tablets
  Other Names: Merck & Co.
  Arms: Pepcid

SUMMARY:
The objective of this study was to compare the single-dose relative bioavailability of Reddy Cheminor and Merck &Co, pepcid 40 mg famotidine tablets under fasting conditions.

DETAILED DESCRIPTION:
Detailed Description : The study was conducted as an open-label, randomized, single-dose, 2-way crossover, relative bioavailability study performed on 30 healthy adult male volunteers. A total of 30 subjects completed the clinical phase of the study. Single oral 40 mg doses were separated by a washout period of 7 days.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

History or presence of significant:

• cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease.

In addition, history or presence of:

* alcoholism or drug abuse within the past year;
* hypersensitivity or idiosyncratic reaction to famotidine or any other histamine H2-receptor antagonist; Subjects who have been on an abnormal diet (for whatever reason) during the four weeks preceding the study.

Subjects who, through completion of the study, would have donated in excess of:

* 500 mL of blood in 14 days, or
* 500 - 750 mL of blood in 14 days (unless approved by the Principal Investigator),
* 1000 mL of blood in 90 days,
* 1250 mL of blood in 120 days,
* 1500 mL of blood in 180 days,
* 2000 mL of blood in 270 days,
* 2500 mL of blood in 1 year. Subjects who have participated in another clinical trial within 28 days of study start.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 1998-10; Primary Completion 1998-10 (Actual); Study Completion 1998-10 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | predose,0. 5, 1, 1. 33, 1. 67, 2, 2. 33, 2.67, 3, 3. 33, 3. 67, 4, 4. 5, 5, 6, 8, 10, 12, 16 and 24 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Serfaty, MD, Principal Investigator — Phoenix Clinical Research Center
Locations (1):
- Phoenix Clinical Research Center, Montreal, Canada